CLINICAL TRIAL: NCT03868917
Title: Comparison of Ultrasound-guided Approach and Ultrasound-guided Approach Combined With Pressure Measurement Technique to Thoracic Paravertebral Block for Open Thoracotomy
Brief Title: Ultrasound-guided Approach Combined With Pressure Measurement Technique to Thoracic Paravertebral Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sangjin Park, professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: apsj07180304
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Thoracotomy

STUDY DESIGN:
Intervention Model Description: Each participant is randomized to one of two groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound group (No Intervention): The participants have continuous thoracic paravertebral block performed using only the ultrasound approach.
- pressure measurement group (Experimental): The participants have continuous thoracic paravertebral block performed using the ultrasound-guided approach combined with pressure measurement techniqueduring needle advancement.
  Interventions: Procedure: thoracic paravertebral block using pressure measurement technique

INTERVENTIONS:
Procedure: thoracic paravertebral block using pressure measurement technique — The continuous thoracic paravertebral block using ultrasound machine is combined with pressure measurement during needle advancement.
  Arms: pressure measurement group

SUMMARY:
Posterolateral thoracotomies are among the most painful procedures of surgery and may cause severe postoperative chest pain and impaired respiratory performance. Paravertebral block (PVB) is an established method of administering postoperative analgesia for thoracic procedures. PVB blocks the somatic and sympathetic nervous systems and is placed by injecting a local anesthetic (LA) into the paravertebral space where the nerve and its branches are located after exiting the intervertebral foramen. But previous study showed 5-10% of failure rate in PVB using ultrasound machine. Pressure measurement during needle advancement could improve reliability of correct needle placement. When the needle tip reaches paravertebral space, there is a sudden lowering of pressures due to respiratory cycle. Therefore, sensitivity and specificity could be improved and correct needle placement become objective and reproducible when PVB using ultrasound is combined with pressure measurement during needle advancement.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective thoracotomy
* ASA status 1,2

Exclusion Criteria:

* Inability to provide adequate informed consent
* Any contraindication to the placement of thoracic paravertebral catheters
* Unstable vertebral and transverse process fractures
* Any chronic painful conditions or preoperative opioid use Any chronic painful conditions or preoperative opioid use
* Coagulation abnormalities or expectation to be on therapeutic anticoagulants postoperatively
* Allergy to any of the drugs/agents used in study protocol
* Altered mental status or emergency surgery
* Comorbid conditions such as sepsis, unstable angina, congestive heart failure

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale for pain (VAS) at 2 hour after the arrival of postanesthetic care unit (PACU) | 2 hour after the arrival of PACU
  VAS score is measured at 2 hour after a patient arrives in PACU. The pain VAS is a unidimensional measure of pain intensity. The pain VAS is a continuous scale comprised of a horizontal (HVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme (no pain 0, maximal pain 100).

CONTACTS AND LOCATIONS:
Overall Officials: SANGJIN PARK, MD, Principal Investigator — Yeungnam University Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yeungnam University hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing is needed to get permission from IRB.

REFERENCES:
- [Result] Syal K, Chandel A. Comparison of the post-operative analgesic effect of paravertebral block, pectoral nerve block and local infiltration in patients undergoing modified radical mastectomy: A randomised double-blind trial. Indian J Anaesth. 2017 Aug;61(8):643-648. doi: 10.4103/ija.IJA_81_17. PMID 28890559
- [Result] Zupcic M, Graf Zupcic S, Duzel V, Simurina T, Sakic L, Fuduric J, Persec J, Milosevic M, Stanec Z, Korusic A, Barisin S. A combination of levobupivacaine and lidocaine for paravertebral block in breast cancer patients undergoing quadrantectomy causes greater hemodynamic oscillations than levobupivacaine alone. Croat Med J. 2017 Aug 31;58(4):270-280. doi: 10.3325/cmj.2017.58.270. PMID 28857520